CLINICAL TRIAL: NCT06683040
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Efficacy and Safety of Oxacom® in Different Dosages in Patients With Pulmonary Arterial Hypertension
Brief Title: Evaluation of the Efficacy and Safety of Oxacom® in Patients With Pulmonary Arterial Hypertension
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXA-PAH-1; ОКСА-ЛАГ-1 (Other: Protocol ID in Cyrillic script)
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Oxaсom; Pulmonary Arterial Hypertension; New Russian drug
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0.030 mg\kg (Experimental)
  Interventions: Drug: Oxacom
- 0.100 mg\kg (Experimental)
  Interventions: Drug: Oxacom
- 0.170 mg\kg (Experimental)
  Interventions: Drug: Oxacom
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxacom — Lyophilisate for solution for intravenous administration, 6.3 mg
  Arms: 0.030 mg\kg; 0.100 mg\kg; 0.170 mg\kg
Drug: Placebo — 0.9% sodium chloride
  Arms: Placebo

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled, phase II-III clinical trial to evaluate the efficacy and safety of the study drug in adult patients with pulmonary arterial hypertension (PAH).

The trial will evaluate the efficacy and safety of both single and multi-dose (seven-day) administrations of the study drug in three dosages: 0.03 mg/kg, 0.10 mg/kg, and 0.17 mg/kg.

The trial is an observer-blinded trial, since the appearance of the study drug and Placebo differs from each other. Patients included in the trial, as well as trial coordinators, investigators, and study center staff will be blinded. The only unblinded staff in the study centers will be those who preparing IP/Placebo and administering IP/Placebo to the study patients.

The trial will include 200 patients with PAH, who will be sequentially included in the trial in two stages.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PAH II or III functional class according to WHO classification
* Symptomatic PAH group 1 according to clinical classification
* Patients who have not previously received any PAH-specific therapy OR patients who have received endothelin receptor antagonists and/or iloprost/selexipag at stable doses for at least 3 months prior to the initial right heart catheterization.
* Ability to perform reproducible 6-min walking test at the screening with a distance from 150 to 450 m.

Exclusion Criteria:

* as per the study protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary vascular resistance (PVR) will be measured to assess and evaluate the efficacy of study drug in comparison with placebo in patients with pulmonary arterial hypertension (PAH). | 6 hours after the start of the IP administration
  To evaluate the efficacy of single doses of the investigational product compared with placebo in patients with pulmonary arterial hypertension (PAH), we will measure pulmonary vascular resistance (PVR)

CONTACTS AND LOCATIONS:
Overall Officials: Tamila V Martynyuk, MD, Principal Investigator — E.I.Chazov Cardiology Center
Locations (1):
- NMCRCardiologyRu, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Russian registry of clinical trials record — https://grlsbase.ru/clinicaltrails/clintrail/13628